CLINICAL TRIAL: NCT06773728
Title: Evaluation of the Impact of Integrating Dynamic Patient-Specific Motion by Implementing Jaw Tracking Systems and Artificial-intelligence Tools in the Attribution of the Occlusion in Full Arch Restorations Through a Digital Workflow: a Clinical Study
Brief Title: Evaluation of the Impact of Integrating Dynamic Patient-Specific Motion and Implementing a Jaw Tracking System in the Attribution of the Occlusion in Full-Arch Restorations Through a Digital Workflow: a Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Panagiotis Ntovas, PhD canditate, National and Kapodistrian University of Athens
Other Study IDs: STUDY0234:
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Jaw Tracking; Occlusion
Keywords: jaw tracking; dental occlusion; artificial intelligence; maxillomandibular position
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Control
  Interventions: Device: Record occlusal contacts; Device: Tracking of jaw movement

INTERVENTIONS:
Device: Record occlusal contacts — Register using a digital device (t-scan) the occlusal contacts
Device: Tracking of jaw movement — An optical jaw tracking system (Modjaw, Modjaw) is going to be implemented
Device: Tracking of jaw movement — Jaw tracking will be performed using an optical jaw tracking system (Zebris, Zebris medical)

SUMMARY:
The maxillomandibular relationship of diagnostic and definitive casts is a fundamental procedure in prosthodontics. Depending on the prosthodontic treatment involvement, different maxillomandibular relationship records can be selected, including maximal intercuspal position (MIP), centric relation (CR) or most comfortable position. Intraoral scanners (IOSs) provide a digital alternative to obtain diagnostic and definitive casts, as well as the maxillomandibular relationship, by acquiring virtual occlusal records.4 Various techniques are available for tracking and recording the mandibular motion of the patient, including mechanical, photographic, radiographic, electromagnetic, ultrasonic-based devices, and optical motion capturing systems. By implementing a digital jaw tracker, patient's individualized mandibular movement can be recorded and combined with intraoral patient's scan, in order to be simulated through the cad software. However, the accuracy of the maxillomandibular relationship has been evaluated only by one study and for one patient. Also, the accuracy to record and replicate of occlusal contacts, acquired by using optical jaw tracking systems has not been evaluated clinically yet. The purpose of the present study was to clinically evaluate the impact of integrating dynamic patient specific-motion and registration, utilizing a digital jaw analyzer (ModJaw), in the attribution of the occlusion.

DETAILED DESCRIPTION:
Patients that are already have been planned for a prosthetic treatment are going to be included in the present research. The records that are used in order to perform an static and a dynamic registration of the occlusion and are standard of care in prosthodontic clinic, will be performed and be obtained by the PI.

In the 1st appointment for each participant a digital impression, as well as a bite registration of the patient will take place in maximal intercuspation(MI) and in the centric relation(CR) implementing am intraoral scanner.(Trios 4, 3Shape).

Patient's individualized dynamic jaw motion will be also recorded by a digital jaw tracking device (ModJaw). In the same appointment patient's contact points will be digitally captured by the scan of the existing teeth or restorations, after the use of an articulating film (8μ , TrollFoil).

Two prototypes utilizing the registration of the jaw tracker in CR and in MCP and two prototypes utilizing the registration that was obtained by the intraoral scanner will be designed. Prototypes will be designed in order to be able to fit over the patient's existing denture.

In the 2nd appointment prototypes will be checked intraorally by implementing an articulating film. An intraoral scan will be performed in order to digitally capture the intraoral markings. Finally patients will be asked to fill out a Visual Analog Scale from 0-100, in order to express "How comfortable they fill their bite, for each one of the prototypes". The questionnaire will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

Patient age ≥ 18 years Patients with ≥ 10 teeth in each dental arch

Exclusion Criteria:

- Patients with a local or systemic conditions contra-indicating dental treatment (hypertension, a heart attack < 1 year, a stroke < 1 year, uncontrolled cardiovascular diseases, uncontrolled diabetes , immunodeficiency, active oral infection as active herpetic lesions etc.) Pregnancy Fully edentulous patients Presence of craniofacial syndromes Patients age <18 Association with an active orofacial trauma

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting the university's clinic
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Occlusal contacts | From the same appointment
  The total number of the true positive and the false positive occlusal contacts between the maxillomandibular relationship obtained from each investigated method is going to be assessed

SECONDARY OUTCOMES:
Patient's acceptance | The visual analog scale records are going to be obtained in the same appointment.
  The mean score for each investigated method, as it will be obtained from the visual analog scale, will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
To further protect patient's data and increase blindness during data analyses

REFERENCES:
- [Background] Revilla-Leon M, Fernandez-Estevan L, Barmak AB, Kois JC, Perez-Barquero JA. Accuracy of the maxillomandibular relationship at centric relation position recorded by using 3 different intraoral scanners with or without an optical jaw tracking system: An in vivo pilot study. J Dent. 2023 May;132:104478. doi: 10.1016/j.jdent.2023.104478. Epub 2023 Mar 6. PMID 36889536
- [Background] Revilla-Leon M, Zeitler JM, Fry E, Kois JC. Digital workflow to measure the mandibular range of motion using different jaw tracking technologies. J Prosthet Dent. 2025 Oct;134(4):1208-1215. doi: 10.1016/j.prosdent.2023.12.018. Epub 2024 Jan 18. PMID 38242763
- [Background] Kois JC, Zeitler JM, Revilla-Leon M. Use of an optical jaw tracking system to capture the envelope of function when designing interim and definitive prostheses: A dental technique. J Prosthet Dent. 2025 Nov;134(5):1472-1479. doi: 10.1016/j.prosdent.2024.03.048. Epub 2024 May 18. PMID 38762385
- [Background] Taut M, Chanteux S, Kui A, Buduru R, Negucioiu M, Manziuc M, Gheorghiu I, Hedesiu M, Buduru S, Ilea A. Condylar Parameters and Mandibular Movement Patterns in Bruxers Using an Optical Jaw Tracking System. J Clin Med. 2024 Dec 19;13(24):7761. doi: 10.3390/jcm13247761. PMID 39768684